CLINICAL TRIAL: NCT06991309
Title: Mindfulness-based Stress Reduction Effects on Depression, Anxiety and Internalized Stigma Compared With Treatment-As-Usual Among Head and Neck Cancer Patients: A Randomized Controlled Trial
Brief Title: Mindfulness-based Stress Reduction Effects on Depression, Anxiety and Internalized Stigma Compared With Treatment-As-Usual Among Head and Neck Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Mohammad Farris Iman Leong Bin Abdullah, Principal investigator, Universiti Sultan Zainal Abidin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LHGJ20230512
Record Dates: First submitted 2025-05-19; First posted 2025-05-27 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Depression, Anxiety; Cancer of the Head and Neck; Psycho-Oncology
Keywords: Depression; Anxiety; Internalized stigma; head and neck cancer; randomized controlled trial
MeSH Terms: conditions — Depression; Anxiety Disorders; Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based stress reduction group (Experimental): MBSR will be conducted as group sessions, with each session lasts for 2.5 hours, once a week for 8 weeks with another 45 minutes of home practice on daily basis.
  Interventions: Behavioral: MBSR
- Treatment-as-usual control group (No Intervention): The participants in the control group will receive treatment-as-usual in which routine oncology support such as appointment with oncologists or palliative care physicians, general practitioner for usual cancer care. The participants physical health and medications for their cancer treatment will be reviewed and treatment will be modified according to physical symptoms such as pain. Specific psychological interventions such as cognitive behavioral therapy, interpersonal therapy, mindfulness-based interventions, acceptance and commitment therapy, etc will be avoided.

INTERVENTIONS:
Behavioral: MBSR — MBSR will be conducted as group sessions, with each session lasts for 2.5 hours, once a week for 8 weeks with another 45 minutes of home practice on daily basis. The MBSR sessions will be based on therapy format developed by Kabat-Zinn. All the sessions focus on mindfulness practices, sharing of experiences with others, and didactic teaching on stress. Mindfulness practices which will be discussed include body scan exercise, and mindful breathing meditation techniques, three-minute breathing exercises, five-minute seeing or hearing exercises, bodily mindfulness in movement and mindful stretching, yoga and sitting meditation. The therapists will review feedbacks for each session, acknowledge the thoughts, feelings, and senses, examine how participants practice mindfulness, and give assignments to encourage participants to continually practice mindfulness at home. Each participant will receive a CD detailing on meditation practices and a workbook on the mindfulness practices.
  Arms: Mindfulness-based stress reduction group

SUMMARY:
Head and neck cancer patients are vulnerable to various psychological complications due to the effects of both cancer itself and cancer treatment on patients' appearance and physical well-being. Nevertheless, few data have been obtained on effective psychosocial interventions that could protect this group of cancer patients' psychological well-being. Therefore, this two-armed, parallel-group, double-blind, randomized control trial (RCT) aims to evaluate and compare the effects of mindfulness-based stress reduction (MBSR) on psychosocial complications (depression, anxiety, and internalized stigma) among newly diagnosed head and neck cancer patients. This RCT will target newly diagnosed head and neck cancer patients who have been treated only with surgery or who have not yet received any treatment. In total, 106 patients who meet all of the study's inclusion criteria and none of its exclusion criteria will be randomly assigned into two groups-an MBSR group and a treatment-as-usual control group-at a 1:1' allocation ratio. Participants in the intervention group (MBSR group) will undergo an eight-week group intervention program. During this program, each intervention will comprise eight modules based on MBSR manual. Outcome assessments will be performed across a three-point timeline, including before the intervention (T0), immediately after the psychosocial intervention at eight weeks (T1), and 12 weeks after the intervention (T2). The primary outcome that will be assessed during this RCT is the severity of depression and anxiety. Meanwhile, the secondary outcome that will be evaluated in this study is such as internalized stigma.

DETAILED DESCRIPTION:
Head and neck cancer differs from other cancer types due to various psychosocial issues associated with it. Moreover, the devastating complications of both cancer itself and cancer treatments' side effects-such as fatigue, pain, speech and swallowing problems, breathing problems, mucositis, xerostomia, and trismus-further disrupt many functions and daily living activities, increasing psychological distress and decreasing QoL. Therefore, an investigation of the psychosocial interventions that could enhance PTG, hope, optimism, and QoL among head and neck cancer patients is crucial. Reducing these patients' internalized stigma and EA could also ultimately restore these cancer survivors' mental and physical well-being. ACT and MBSR have been reported to enhance positive psychology and alleviate psychological distress among cancer patients. However, data regarding ACT and MBSR's effects on positive psychology, psychological sequelae and QoL in head and neck cancer patients are lacking. ACT's effects on PTG, hope, optimism, QoL, depression, anxiety, and EA among head and neck cancer patients have not been studied. Although MBSR has been reported to lower psychological distress and enhance QoL in head and neck cancer patients, its effects on positive psychology and EA have not been investigated. Hence, MBSR may act as a good comparator intervention to ACT for evaluating its efficacy on positive psychology, psychological sequelae and QoL among head and neck cancer patients. Therefore, we have proposed a three-armed RCT to evaluate these effects over time compared to a control group receiving treatment-as-usual.

Objectives:

Primary objectives:

Evaluate MBSR's efficacy in alleviating the severity of depression and anxiety among head and neck cancer patients compared to a control (treatment-as-usual) immediately after the eight-week intervention and 12 weeks post-intervention compared to pre-intervention.

Secondary objective:

Examine MBSR's efficacy in alleviating internalized stigma among head and neck cancer patients compared to a control (treatment-as-usual) immediately after the eight-week intervention and 12 weeks post-intervention compared to pre-intervention.

Methods/design:

Design:

The current study will conduct a multicentre, two-armed, parallel-group, double-blind RCT that conducted over one and a half year.

Setting This study will be conducted in Advanced Medical and Dental Institute (AMDI) at the Universiti Sains Malaysia (USM) and Universiti Kebangsaan Malaysia Medical Centre (UKMMC).

Support and ethics This study has received approval from the Human Research Ethics Committee of Universiti Sains Malaysia (code: USM/JEPeM/21040336). The study will be conducted in compliance with the Declaration of Helsinki (1974) and its amendments, as well as the Malaysian Good Clinical Practice Guidelines for Clinical Trials. The institutional review board will be informed of any modification to the study's protocol (such as its eligibility criteria, study procedures, outcome measures, scheduled interventions, and data analyses) in writing. This manuscript was written without any deviation from the original protocol submitted to the Human Research Ethics Committee of Universiti Sains Malaysia.

The principal investigator will lead the trial center and closely coordinate with the research coordinator and the site coordinator, participate in subject recruitment, and oversee the study's consent procedures. A trial monitoring committee has been established.

All participants will be permitted to withdraw from the study at any time without specifying the reason for their withdrawal, and we will not use any of the information collected from participants who choose to withdraw. Prior to their participation in this study, participants will be informed that the results of this study will only be used for research purposes and will not be recorded in patients' case files. Participants' personally identifiable information will not be sought or recorded, and participants' anonymity will be assured. Each participant will be sequentially assigned a research number (e.g., RCT001, RCT002, etc.). All documents involved in this study's assessment of research subjects-including participants' personal information (socio-demographic, substance history, symptomatology, and questionnaire responses)-will be stored in document files and locked in a cabinet whose key is kept by the corresponding author.

Participants may also withdraw from the study if an adverse event occurs. An adverse event (AE) is any untoward medical occurrence involving a participant in a trial intervention that does not necessarily causally relate to this treatment. An AE can be any unfavorable or unintended sign, symptom, or disease that is temporarily associated with the use of an investigational intervention, whether related or unrelated to the investigational intervention. Participants will be issued a study card featuring the research team's contact details and encouraged to maintain close contact by phone and report any AE.

If an unexpectedly serious AE is reported in a subject or more in any of the randomized intervention group (MBSR), an interim analysis will be conducted to investigate this matter. If the findings of this investigation indicate any safety concerns which is related to the intervention administered (MBSR), the Trial Monitoring Committee will terminate the trial prematurely. Serious AE which are indication for premature termination of trial include suicidal tendency, life-threatening self-harm, and hospitalization related to psychological adverse events arise from the intervention administered.

Only the study's corresponding author and co-authors are permitted to access the study's files for data analysis or publication purposes. The findings of this study will be submitted for publication in peer-reviewed academic journals and for presentation at international conferences and symposia. The study's principal investigator will be listed as the corresponding author, and authorship eligibility will be based on the International Committee of Medical Journal Editors' recommendations.

All of this study's investigators declare no financial or other competing interests in conducting this study.

Participants:

This study's participants will be recruited from the source population. This population includes all newly diagnosed head and neck cancer patients who have been treated only with surgery or who have not yet received treatment and who are registered under the oncology and otorhinolaryngology unit of the Advanced Medical and Dental Institute (AMDI) at the Universiti Sains Malaysia (USM) or the oncology and otorhinolaryngology unit of Universiti Kebangsaan Malaysia Medical Centre (UKMMC). The sample size was estimated using the sample size calculator developed by Lu et al. (2008) for mixed linear models. Key parameters included a standard mean difference of 0.65, a type I error of 0.05, power of 0.8, a 1:1 group allocation ratio, three time points, and estimated attrition rates of 10% (from T0 to T1) and 20% (from T1 to T2). Based on these calculations, the estimated sample size was 53 participants per group.

Recruitment process:

This study will use a consecutive sampling method. The research team will approach head and neck cancer patients registered at the two targeted institutions and explain the study's objectives and procedures. Patients who are interested in participating in this study will be screened for inclusion and exclusion criteria by a research team member. All eligible patients will be invited to participate in this study. The study's purposes and procedures will be thoroughly explained (verbal explanation by the research assistant and a copy of the participant information will also be distributed) to prospective participants before they are invited to participate in this study, their anonymity will be assured, and they will be informed of their right to withdraw from the study at any time and the data collected will be discarded. Eligible patients will be given 48 hours to decide on their participation in the study. Then, participants will sign written informed consent to participate in the study before they enroll in the study.

Randomization:

This study will use stratified permuted block randomization, stratifying trial participants according to their age (18 to 40 years old, 41 to 60 years old, and over 60 years old) and gender (male and female). Participants will be randomized into two groups: an MBSR group and a control group of patients on treatment-as-usual for intervention. Using a 1:1 allocation ratio and block randomization, we will randomly assign participants to the two groups. An allocation sequence will be generated via computer-generated random numbers, which will be obtained by a research assistant who is not otherwise involved in this study. The allocation sequence will be concealed in an opaque, sequentially numbered envelope.

Interventions:

An eight-week psychosocial intervention will be administered to participants in the intervention group (MBSR) while participants in the control group will receive treatment-as-usual. The study's outcomes will be assessed at three times: pre-intervention (T0), immediately after the eight-week intervention (T1), and 12 weeks after the intervention (T2).

The MBSR intervention will comprise eight sessions delivered at a rate of one session per week. Each session will last for 2.5 hours. At AMDI, USM, and UKMMC, chemotherapy for head and neck cancer lasts for 8 weeks, delivered at a rate of one session per week. Similarly, radiotherapy for head and neck cancer lasts for eight weeks at these institutions. Therefore, this study's MBSR sessions will align with participants' chemotherapy or radiotherapy sessions to ensure that all participants attend their intervention sessions. MBSR will be provided in group settings with intervention groups of 10 participants each.

Mindfulness-based stress reduction (MBSR):

MBSR will be conducted as group sessions, with each session lasts for 2.5 hours, once a week for 8 weeks with another 45 minutes of home practice on daily basis. The MBSR sessions will be based on therapy format developed by Kabat-Zinn. All the sessions focus on mindfulness practices, sharing of experiences with others, and didactic teaching on stress. Mindfulness practices which will be discussed include body scan exercise, and mindful breathing meditation techniques, three-minute breathing exercises, five-minute seeing or hearing exercises, bodily mindfulness in movement and mindful stretching, yoga and sitting meditation. The therapists will review feedbacks for each session, acknowledge the thoughts, feelings, and senses, examine how participants practice mindfulness, and give assignments to encourage participants to continually practice mindfulness at home. Each participant will receive a CD detailing on meditation practices and a workbook on the mindfulness practices.

Treatment-as-usual control group:

The participants in the control group will receive treatment-as-usual in which routine oncology support such as appointment with oncologists or palliative care physicians, general practitioner for usual cancer care. The participants physical health and medications for their cancer treatment will be reviewed and treatment will be modified according to physical symptoms such as pain. Specific psychological interventions such as cognitive behavioral therapy, interpersonal therapy, mindfulness-based interventions, acceptance and commitment therapy, etc will be avoided.

Treatment fidelity:

MBSR will be conducted for the MBSR group by a therapist trained in MBSR, and a trained backup therapist will be on standby to replace the primary therapist when necessary. All the study's therapists and backup therapists will be postgraduate students in psychology who are not otherwise involved in the study. All the therapists have two-year experience of conducting psychotherapy. They will also receive training manual detailing the psychotherapy sessions for MBSR.

Blinding:

The researchers will also be "blinded" for the study since the participants' randomized assignment into the designated groups will be conducted by a research assistant who is not otherwise involved in the study or data analysis. This project's data collection will also be conducted by that research assistant who is not otherwise involved in the study or data analysis and who is unaware of the study's hypotheses. Moreover, the project's data analysis will be conducted by statisticians who are not otherwise involved in the study. A statistical analysis plan is established prior to the final unblinded of the data lock.

Measures:

Data collection will be conducted every weekday during working hours, and flyers announcing the study and the benefits of participating in this study will be disseminated to all newly diagnosed head and neck cancer patients at the study's focal institutions (within one month of their diagnosis) in order to ensure adequate subject enrolment to achieve the calculated sample size. This clinical trial protocol was written according to the CONSORT 2025 Statement: updated guideline for reporting randomised trials.

Sociodemographic and tumor characteristics:

The sociodemographic characteristics which will be recorded from each participant include age, gender, ethnicity, marital status, education, and employment status. While the tumor characteristics which will be gathered from the participants are duration of cancer diagnosis, types of head and neck cancer, stage of cancer and modalities of cancer treatment received.

Primary outcomes:

Depression and anxiety: The Malay version of the "Hospital Anxiety and Depression Scale" (HADS) will be used to assess the severity of depression and anxiety symptoms among participants.

Secondary outcome:

Internalized stigma: The Malay version of the "Shame and Stigma Scale" (SSS) will be used to measure the degree of internalized stigma among participants.

Other measures:

The participants compliance to the interventions will be recorded as they will be requested to fill in electronic dairies regarding their performance of the home assignments and practice of the interventions at home. The reasons for absence from therapy sessions, dropouts and loss to follow up (such as loss of interest to participate, dislike of the intervention, not feeling well or death) will also be recorded.

Data analysis:

All of this study's data analysis will be conducted using the Statistical Package for Social Sciences, version 26. Initially, the baseline sociodemographic and tumor characteristics will be presented by randomized groups (MBSR and control groups).

The mean difference in the primary outcome (HADS score) for the two randomized groups (MBSR and control groups) at each specific time point (pre-intervention [t0], post-treatment at 8 weeks [t1] and 12 weeks after intervention [t2]) will be assessed using mixed linear model will be employed for comparing the primary outcomes (HADS- Depression and Anxiety Subscores) between between MBSR and control groups across the three time points (t0, t1 and t2), while controlling for stratification factors such as age and gender. The main effects of intervention in the groups and time points will be presented as standardized mean difference. The study's primary analysis will follow the intention-to-treat (ITT) principle. The data analysis for the study's secondary outcome (total SSS score) will be conducted similarly to the primary outcomes' calculation. In addition, 95% confidence interval will also be presented alongside the main effect. Statistical significance will be two-tailed and set to p < 0.05. Missing data will be handled accordingly.

ELIGIBILITY:
Inclusion Criteria:

* those diagnosed with HNC confirmed by histopathological report and at any stage of cancer
* those aged 18 years old and above
* those who have completed surgery and started chemotherapy and/or radiotherapy
* literate in the Malay language.

Exclusion Criteria:

* history of pre-existing psychiatric illnesses (such as psychotic disorder, bipolar disorder, anxiety disorder, depressive disorder, neurodevelopmental disorder, neurocognitive disorder)
* history of pre-existing medical illnesses which may induce psychiatric symptoms (such as kidney and liver failure, ischemic heart disease, epilepsy, hyperthyroidism, hypothyroidism, Cushing's syndrome, Addison's disease, systemic lupus erythematosus, neurological disorder, rheumatoid arthritis)
* history of illicit drug and alcohol use
* pregnancy
* suicidal tendency
* those with history of engaged in other psychotherapy
* those who are not physically and cognitively fit to participate in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale | Change of the mean HADS Depression and Anxiety Subscale scores between baseline and 8 weeks of commence of intervention and between 8 weeks of commence of intervention to 12 weeks after completion of intervention
  The Malay version of the "Hospital Anxiety and Depression Scale" (HADS) will be used to assess the severity of depression and anxiety symptoms among participants. The HADS is a 14-item, self-rated questionnaire with seven items in each of its subscales. Each item is scored from 0 to 3, and the total score for both the depression and anxiety subscales ranges from 0 to 21 per subscale. The cut-off for depression cases is 8/21, and the cut-off for anxiety cases is also 8/21. The Malay version of the HADS has been validated among Malaysian breast cancer patients, and it exhibited acceptable to good internal consistency for its total score and subscales with Cronbach's alphas ranging from 0.73 to 0.87

SECONDARY OUTCOMES:
Shame and Stigma Scale | Change of the mean total SSS scores between baseline and 8 weeks of commence of intervention and between 8 weeks of commence of intervention to 12 weeks after completion of intervention
  The Shame and Stigma Scale (SSS) is a self-administered instrument employed to measure the degree of internalized stigma of living with cancer among the participants in this study. It consists of 20 items and made up of four domains (shame of appearance, speech and social concerns, sense of stigma and regret). Each item is scored in a Likert scale ranging from 0 (never) to 4 (all the time). Hence, the higher the score, the greater is the degree of internalized stigma. The SSS exhibits good psychometric properties with an excellent internal consistency (Cronbach's α = 0.94). It was translated and validated in the Malay language among the cancer patients population in Malaysia and demonstrated good internal consistency with Cronbach's α of 0.88

CONTACTS AND LOCATIONS:
Locations (1):
- Pusat Perubatan Universiti Sains Malaysia Bertam, Kepala Batas, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No
Study subjects are vulnerable group of the population and restriction of IPD is part of the requirement of the institutional review board to protect the personal data of the subjects.

REFERENCES:
- [Derived] Zhang Z, Zhang Q, Lu P, Shari NI, Nik Jaafar NR, Mohamad Yunus MR, Qiu Q, Ismail F, Ab Muin NF, Leong Bin Abdullah MFI. Mindfulness-Based Stress Reduction Alleviates Depression, Anxiety, and Internalized Stigma Compared With Treatment-as-Usual Among Head and Neck Cancer Patients: Findings From a Randomized Controlled Trial. Depress Anxiety. 2025 Sep 11;2025:7499120. doi: 10.1155/da/7499120. eCollection 2025. PMID 40979247